CLINICAL TRIAL: NCT00430846
Title: A Phase I Dose Escalation Study of SGN-35 in Patients With Relapsed/Refractory CD30-Positive Hematologic Malignancies.
Brief Title: Phase I Open-Label Dose Finding Study of SGN-35 for CD30 Positive Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG035-0001; NCT00412282 (obsolete NCT alias)
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Lymphoma, Non-Hodgkin; Disease, Hodgkin; Lymphoma, Large-Cell, Anaplastic
Keywords: Antigens,CD30; Antibody-Drug Conjugate; Antibodies, Monoclonal; Lymphoma, Non-Hodgkin; Disease, Hodgkin; Lymphoma, Large-Cell, Anaplastic; Hematologic Diseases; Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Hematologic Diseases; Lymphoma | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: SGN-35

INTERVENTIONS:
Drug: SGN-35 — Every 21 days. Dose Escalating. 0.1 - 3.6 mg/kg
  Other Names: brentuximab vedotin

SUMMARY:
Phase I study to define the safety profile and pharmacokinetic parameters of SGN-35 in patients with relapsed/refractory CD30-positive hematologic malignancies. This is a single-arm, open-label, Phase I dose escalation study designed to define the MTD, PK, immunogenicity and anti-tumor activity of SGN-35 in patients with relapsed/refractory CD30-positive hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed CD30-positive hematologic malignancy.
* Patients with HL must have failed systemic chemotherapy either as induction therapy for advanced stage disease or salvage therapy after initial radiotherapy for early stage disease and were ineligible for, refused treatment by, or previously received stem cell transplant.
* Patients must have measurable disease of at least 10mm as documented by radiographic technique.
* Must be at least 18 years of age.

Exclusion Criteria:

* Patients with current diagnosis of pcALCL (systemic ALCL eligible).
* Patients with history of allogeneic stem cell transplant.
* Patients who have had previous treatment with any anti-CD30 antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events and laboratory abnormalities | 1 month after last dose

SECONDARY OUTCOMES:
PK profile | 2 months after last dose
Immunogenicity (anti-SGN-35 antibodies) | 1 month after last dose
Anti-tumor activity | 1 month after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Andres Forero, MD, Principal Investigator — University of Alabama at Birmingham; Anas Younes, MD, Principal Investigator — M.D. Anderson Cancer Center; Nancy Bartlett, MD, Principal Investigator — Washington University School of Medicine; John Leonard, MD, Principal Investigator — Weill Medical College of Cornell University; Dana Kennedy, PharmD, Study Director — Seagen Inc.
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Washington University, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - University of Texas/MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Younes A, Bartlett NL, Leonard JP, Kennedy DA, Lynch CM, Sievers EL, Forero-Torres A. Brentuximab vedotin (SGN-35) for relapsed CD30-positive lymphomas. N Engl J Med. 2010 Nov 4;363(19):1812-21. doi: 10.1056/NEJMoa1002965. PMID 21047225
- [Derived] Suri A, Mould DR, Song G, Kinley J, Venkatakrishnan K. Population Pharmacokinetics of Brentuximab Vedotin in Adult and Pediatric Patients With Relapsed/Refractory Hematologic Malignancies: Model-Informed Hypothesis Generation for Pediatric Dosing Regimens. J Clin Pharmacol. 2020 Dec;60(12):1585-1597. doi: 10.1002/jcph.1682. Epub 2020 Jun 28. PMID 32596842